CLINICAL TRIAL: NCT04729010
Title: Acupuncture as a Symptomatic Treatment for Anxiety in Parkinson's Disease
Brief Title: Acupuncture for Anxiety in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, Kim Yun Jin, Associate Professor, Xiamen University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITCM0005
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Anxiety
Keywords: Acupuncture, Anxiety, Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Subjects receive a sham acupuncture. (Sham Comparator): Subjects will be randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Interventions: Other: Acupuncture to treat anxiety in Parkinson disease
- Randomized Subjects receive a real acupuncture. (Active Comparator): Subjects will be randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Interventions: Other: Acupuncture to treat anxiety in Parkinson disease

INTERVENTIONS:
Other: Acupuncture to treat anxiety in Parkinson disease — Subjects will be randomized in a 1:1 ratio to receive sham acupuncture.

SUMMARY:
This is a single-center, double-blind, placebo-controlled trial to see if acupuncture can safely and effectively manage anxiety in Parkinson's Disease. Eligible subjects will receive either real or sham acupuncture THREE times weekly for a total of SIX weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's Disease by authorized Neurologist.
* Patients 40-75 years of age
* Patients who have significant anxiety symptom
* Patients must be on a stable medication regimen for the treatment of PD

Exclusion Criteria:

* Patients who have had previous acupuncture within the past SIX months
* Patients with dementia, depression, or sleep disorder
* Patients who are currently taking medications known to affect anxiety

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Anxiety Scale (HAM-A) between the treatment group. | SIX weeks
  The primary outcome measure will be the change between the baseline visit and the SIX-week time point in the Hamilton Anxiety Scale (HAM-A) between the treatment group. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
Change in the Generalized Anxiety Disorder 7-Item (GAD-7) scale between the treatment group. | SIX Weeks
  The primary outcome measure will be the change between the baseline visit and the SIX-week time point in the Generalized Anxiety Disorder 7-Item (GAD-7) scale between the treatment group. Each item is scored on a scale of 0 (not at all) to 3 (Nearly Every Day), with a total score range of 0-56, where <4 indicates Minimal Anxiety, 5-9 Mild Anxiety, 10-14 Moderate Anxiety, and 15-21 Severe Anxiety.

SECONDARY OUTCOMES:
Change in the Unified Parkinson's Disease Rating Scale between the treatment group. | THREE months
  A comprehensive assessment of both motor and non-motor symptoms associated with Parkinson's. The Unified Parkinson's Disease Rating Scale is made up of 42 items. These items are divided into six sections which are separately "evaluation of mentation, behavior, and mood", "self-evaluation of the activities of daily life", "clinician-scored monitored motor evaluation", "complications of therapy", "Hoehn and Yahr staging of severity of Parkinson's disease" and "Schwab and England ADL scale". The evaluation score for the first item to the 39th item is 0 to 4 points. The evaluation score for the 40th to the 42th item is 0 to 1 points. The higher score means the worse condition. This scores indicate severe symptoms.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR